CLINICAL TRIAL: NCT01857960
Title: Survey About Knowledge and Attitudes Regarding Acne in Mexican Adolescents
Brief Title: Attitudes and Knowledge of Acne in Mexican Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo-Cazares, Dermatology Research Director, Universidad Autonoma de San Luis Potosí
Other Study IDs: AcKNOW
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Acne
Keywords: Acne; Treatment; Cost; Behavior
MeSH Terms: conditions — Acne Vulgaris; Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adolescents: Acne survey among Mexican adolescents
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — A survey is directly applied to subjects who meet the inclusion and exclusion criteria

SUMMARY:
Acne is a chronic inflammatory disease that affects almost 100% of the teenagers worldwide. The peak incidence is between 12 and 18 years old, although it can be present in adults. There are many different beliefs about what can cause or exacerbate acne, and also about treatment.

In Mexico, 26.4% of the population is between 15 and 29 years old, which represents that more than 25% of the population is at risk for presenting acne. In our country, the different beliefs about the causes and treatment of acne among general adolescent population have not been explored. The objective of the present study is to determine the possible causes for which young Mexicans do not go to the dermatologist to receive treatment for acne. Our main hypothesis is that the lack of knowledge of the disease is responsible for this behavior.

DETAILED DESCRIPTION:
Acne is a chronic inflammatory disease that affects almost 100% of the teenagers worldwide. The peak incidence is between 12 and 18 years old, although it can be present in adults. There are many different beliefs about what factors can cause or exacerbate acne, as well concerning treatments.

In Mexico, 26.4% of the population is between 15 and 29 years old, which represents that more than 25% of the population is at risk for presenting acne. In our country, there are diverse beliefs about the causes and treatment of acne among general adolescent population which have not been explored before. The objective of the present study is to determine possible causes that are involved in the low use of health system with the intention to receive treatment for acne. The investigators' main hypothesis is that the lack of knowledge of the disease is responsible for this behavior.

The investigators are going to explore health, educational, family and economic issues in the search of association by multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Mexican subjects
* Age between 12 and 25 years
* Both genders
* Sign informed consent

Exclusion Criteria:

* None

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Community high schools and colleges.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-01 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Cause for not receiving medical treatment | Up to 1 year
  To determine the possible causes for which an adolescent does not look for medical treatment for acne

SECONDARY OUTCOMES:
Description of knowledge about acne | Up to 1 year
  To describe the knowledge that young subjects have regarding the causes of acne
Treatments for acne used by teenagers | Up to 1 year
  To describe the most used treatments for acne among teenagers
Professional indicated to treat acne | Up to 1 year
  To know which professionals (health-care related or not) are considered appropriate by teenagers to treat acne

CONTACTS AND LOCATIONS:
Overall Officials: Bertha Torres-Alvarez, MD, Study Chair — Universidad Autonoma de San Luis Potosi; Juan P Castanedo-Cazares, MD, Study Director — Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Cheng CE, Irwin B, Mauriello D, Liang L, Pappert A, Kimball AB. Self-reported acne severity, treatment, and belief patterns across multiple racial and ethnic groups in adolescent students. Pediatr Dermatol. 2010 Sep-Oct;27(5):446-52. doi: 10.1111/j.1525-1470.2010.01286.x. Epub 2010 Aug 26. PMID 20796234
- [Background] Al Robaee AA. Prevalence, knowledge, beliefs and psychosocial impact of acne in University students in Central Saudi Arabia. Saudi Med J. 2005 Dec;26(12):1958-61. PMID 16380781
- [Background] Smithard A, Glazebrook C, Williams HC. Acne prevalence, knowledge about acne and psychological morbidity in mid-adolescence: a community-based study. Br J Dermatol. 2001 Aug;145(2):274-9. doi: 10.1046/j.1365-2133.2001.04346.x. PMID 11531791